CLINICAL TRIAL: NCT01360346
Title: Multicentric, Single Blind, Randomized Controlled Trial on Enteral Sedation Versus Intravenous Sedation in Critically Ill High-risk ICU Patients
Brief Title: Enteral Versus Intravenous Sedation in Critically Ill High-risk ICU Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Milan (Other)
Collaborators: Ospedale San Paolo (Other); Ospedale Maggiore Policlinico Mangiagalli e Regina Elena (Other); Azienda Ospedaliera San Gerardo di Monza (Other); Azienda Ospedaliera Niguarda Cà Granda (Other); Azienda Ospedaliera Fatebenefratelli e Oftalmico (Other); Fondazione IRCCS Policlinico San Matteo di Pavia (Other); San Luigi Gonzaga Hospital (Other); Ospedale S. Giovanni Bosco (Other); Ospedale Cardinal Massaia (Other); Azienda Ospedaliera, Ospedale Civile di Legnano (Other); Nuovo Ospedale Civile S.Agostino Estense (Other)
Responsible Party: Principal Investigator, Giovanni Mistraletti, University Researcher, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SedaENvsIV
Record Dates: First submitted 2011-05-20; First posted 2011-05-25 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Critical Illness; Mechanical Ventilation Complication
Keywords: Enteral Sedation; Intravenous Sedation; Critically ill ICU patient; Conscious Sedation; Deep Sedation; RASS; CAM-ICU; VNR; BPS; Propofol; Midazolam; Hydroxyzine; Lorazepam; Melatonin
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enteral Sedation (EN) (Experimental): Melatonin, Hydroxyzine, and Lorazepam. At every work shift, it will be checked the possibility to decrease the Lorazepam and then the Hydroxyzine dosage to quickly obtain and continuously maintain a RASS level = 0
  Interventions: Procedure: Enteral Sedation (EN)
- Intravenous Sedation (IV) (Active Comparator): Intravenous propofol or midazolam administration at the ICU admission to discharge at the compatible lowest level with harsh ICU environment. At every shift nurses are requested to give intravenous lowest dosage to obtain RASS=0
  Interventions: Procedure: Control group: Intravenous Sedation (IV)

INTERVENTIONS:
Procedure: Enteral Sedation (EN) — Intravenous propofol or midazolam administration at the ICU admission and stopped within 48h. Melatonin by enteral route (3mg x 2/die) from admission to discharge. Hydroxyzine by enteral route from ICU admission (600mg/die), decreased and stopped as soon as possible. Lorazepam supplementation (maximum 16mg/die) if hydroxyzine is inadequate.
  Other Names: ENTERAL
  Arms: Enteral Sedation (EN)
Procedure: Control group: Intravenous Sedation (IV) — Propofol or midazolam from ICU admission to discharge at the compatible lowest level with harsh ICU environment.
  Other Names: INTRAVENOUS
  Arms: Intravenous Sedation (IV)

SUMMARY:
Recent studies suggest the employment of 'conscious' sedation (1) for critically high - risk patients (2), showing more efficacy then deep sedation (3). The investigators want to compare intravenous injection versus enteral sedative drugs administration, purposing to maintain a 'conscious' sedation level compatibly with the needed cares, invasive procedures, and medical and nursing surveillance.

DETAILED DESCRIPTION:
Recent studies suggest the employment of 'conscious' sedation for critically high - risk patients (2), showing more efficacy then deep sedation (3). From this point of view it's important to consider both the choice of sedative drugs and the way to administer them to maintain the constant 'conscious' sedation level that the investigators wanted.

This research compares two different procedures for sedation therapy: through a randomized and blind controlled trial the interventional group will collect patients receiving sedatives from enteral way (4, 5, 6). In the control arm, sedation administration forecasts intravenous injection (7), recognised like the best practice in the most of intensive care units of the world.

To consider two different clinical approach for administration the investigators have to use different molecules: in the control arm propofol and midazolam will be continuously administered through intravenous injection with daily suspension (7); in the intervention arm the investigators will administer melatonin like a physiological hypnotic inductor (6), the continuous 'conscious' sedation will be maintained through hydroxyzine and eventually lorazepam (4), and all the active principles will be given by enteral administration.

The goal of the study is to compare intravenous injection versus enteral sedative drugs administration, analysing their efficacy and the feasibility to maintain constant the appropriate sedation level (RASS measured = RASS wished ±1) (8) in high - risk patients admitted in Intensive Care Unit (2), purposing to conserve a 'conscious' sedation level compatibly with the needed cares, invasive procedures, and medical and nursing surveillance.

MATERIALS AND METHODS Prospective, randomized and controlled multicentric, single blind trial. Participant ICU centres: San Paolo MI (Iapichino), Policlinico MI (Gattinoni) , Fatebenefratelli MI (Cigada), Niguarda MI (De Gasperi), Desio (Ronzoni), Legnano (Radrizzani), Monza (Pesenti), Belluno (Mazzon), Lugano (Malacrida), Modena (Rambaldi), Torino (Livigni), Asti (Cardellino).

PROCEDURE Bare minimum sedation drug titration will be done to maintain and to achieve prematurely a 'conscious' sedation level (RASS=0). During every shift it will be discussed the appropriate sedation therapy: if physicians choose a deep sedation goal (RASS <-3) this decision has to be explained and registered; then enteral sedation has to be maximized in randomized enteral patients group. If necessary intravenous sedation has to be added , and this procedure dose not represent a violation of research protocol.

If there is pain (VNR>3 or BPS>6) it will be administrated analgesic therapy according to hospital guidelines bare minimum duration. The treatment of procedural pain will be applied both groups trough Fentanest/Morphine + propofol/midazolam bolus intravenous, this procedure dose not represent a violation of research protocol.

If acute cerebral malfunction appears (CAM-ICU positive), it will be administrated haloperidol (1mg per os, max 10 mg/die) or other antipsychotic therapy according to hospital guidelines.

Enteral artificial nutrition with prokinetics will be started as soon as possible both group, while parenteral nutrition will be administered only if strictly necessary. If gastric stagnation > 200 ml/4 hours exceeds 2 days duration, it could be positioned nasogastric tube or digiunostomy.

All patients will be sit in a semiortopnoic position (bed back rest inclination between 30 and 45°).

STUDY POWER AND STATISTICAL ANALYSIS The investigators suppose to obtain a difference of 15% per cent between two arms for patients' sedation adequacy benefit (RASS = desired RASS + 1). Knowing that the enteral approach reached 83% adequacy from a observational monocentric research (5), it should be necessary to enrol 141 patients for each arm (power 80%). In consideration of the missing data, the investigators expect to enroll 300 patients. An "ad interim" statistical analysis is planned after the enrollment of 70 patients in each group.

To provide a statistical analysis as "Intention To Treat" for possible arms change risk.

It's planned to obtain a selective analysis involving each hospital included in the study.

It's planned to obtain a selective analysis about septic patients (greater delirium prevalence) (9).

It's planned to obtain a selective analysis divided for age (greater delirium prevalence if age >70) (10).

The randomization will be achieved trough out a particular Internet Website with a specific program expressly built. It will be used minimization technique to maintain groups balanced in the patients' sample of each centre.

ELIGIBILITY:
Inclusion Criteria:

* High Risk Patients (Ventilation days assessment >3, SAPS II >32).
* Until 24 h after ICU admission
* Age > 18 years

Exclusion Criteria:

* Neurosurgical patients
* Allergy to medications used in the study
* CNS diseases (epilepsy, ictus, dementia, anoxic coma…)
* Liver encephalopathy (Child C)
* Previous psychiatric or cognitive pathology
* Absolute contraindications to use enteral route (acceptable NGT, digiunostomy, ileostomy)
* Pregnant patients or in breast-feeding
* DNR patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-10 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Percent of efficacy, measured by observed RASS = desired RASS ± 1. | One year

SECONDARY OUTCOMES:
Sedation protocol effectiveness: percentage of "protocol violation days" on the total of ICU days. | One year
Delirium and coma free days (respectively negative CAM-ICU and RASS > - 3 in all daily observations until 28° ICU day) (11) | One year
Ventilation free days (12) | One year
Nursing evaluation of sedation adequacy (communication skills, cooperation, environment tolerance) (13) | One year
Overall ICU and hospital mortality, absolute mortality after 1 year from ICU discharge. | 24 months
Sedative drugs costs. | One year
Indirect inefficacy markers | One year
  1. Prevalence of 'dangerous episodes': self - extubation, removal of other invasive clinical instruments;
  2. Length of ICU and hospital stay
  3. Use of anti-psychotic drugs (indirect delirium marker)
  4. Other indicators of sedation failure: use of restraining therapies, antagonist administrations (fluamzenil - naloxone).

CONTACTS AND LOCATIONS:
Overall Officials: Iapichino Gaetano, MD, Study Chair — University of Milan
Locations (1):
- AO San Paolo - Polo Universitario, Milan, Italy

REFERENCES:
- [Background] Strom T, Martinussen T, Toft P. A protocol of no sedation for critically ill patients receiving mechanical ventilation: a randomised trial. Lancet. 2010 Feb 6;375(9713):475-80. doi: 10.1016/S0140-6736(09)62072-9. Epub 2010 Jan 29. PMID 20116842
- [Background] Iapichino G, Mistraletti G, Corbella D, Bassi G, Borotto E, Miranda DR, Morabito A. Scoring system for the selection of high-risk patients in the intensive care unit. Crit Care Med. 2006 Apr;34(4):1039-43. doi: 10.1097/01.CCM.0000206286.19444.40. PMID 16484895
- [Background] Payen JF, Chanques G, Mantz J, Hercule C, Auriant I, Leguillou JL, Binhas M, Genty C, Rolland C, Bosson JL. Current practices in sedation and analgesia for mechanically ventilated critically ill patients: a prospective multicenter patient-based study. Anesthesiology. 2007 Apr;106(4):687-95; quiz 891-2. doi: 10.1097/01.anes.0000264747.09017.da. PMID 17413906
- [Background] Cigada M, Pezzi A, Di Mauro P, Marzorati S, Noto A, Valdambrini F, Zaniboni M, Astori M, Iapichino G. Sedation in the critically ill ventilated patient: possible role of enteral drugs. Intensive Care Med. 2005 Mar;31(3):482-6. doi: 10.1007/s00134-005-2559-7. Epub 2005 Feb 16. PMID 15714324
- [Background] Cigada M, Corbella D, Mistraletti G, Forster CR, Tommasino C, Morabito A, Iapichino G. Conscious sedation in the critically ill ventilated patient. J Crit Care. 2008 Sep;23(3):349-53. doi: 10.1016/j.jcrc.2007.04.003. Epub 2007 Jul 5. PMID 18725039
- [Background] Mistraletti G, Sabbatini G, Taverna M, Figini MA, Umbrello M, Magni P, Ruscica M, Dozio E, Esposti R, DeMartini G, Fraschini F, Rezzani R, Reiter RJ, Iapichino G. Pharmacokinetics of orally administered melatonin in critically ill patients. J Pineal Res. 2010 Mar;48(2):142-7. doi: 10.1111/j.1600-079X.2009.00737.x. Epub 2010 Jan 8. PMID 20070489
- [Background] Girard TD, Kress JP, Fuchs BD, Thomason JW, Schweickert WD, Pun BT, Taichman DB, Dunn JG, Pohlman AS, Kinniry PA, Jackson JC, Canonico AE, Light RW, Shintani AK, Thompson JL, Gordon SM, Hall JB, Dittus RS, Bernard GR, Ely EW. Efficacy and safety of a paired sedation and ventilator weaning protocol for mechanically ventilated patients in intensive care (Awakening and Breathing Controlled trial): a randomised controlled trial. Lancet. 2008 Jan 12;371(9607):126-34. doi: 10.1016/S0140-6736(08)60105-1. PMID 18191684
- [Background] Sessler CN, Gosnell MS, Grap MJ, Brophy GM, O'Neal PV, Keane KA, Tesoro EP, Elswick RK. The Richmond Agitation-Sedation Scale: validity and reliability in adult intensive care unit patients. Am J Respir Crit Care Med. 2002 Nov 15;166(10):1338-44. doi: 10.1164/rccm.2107138. PMID 12421743
- [Background] Pandharipande PP, Sanders RD, Girard TD, McGrane S, Thompson JL, Shintani AK, Herr DL, Maze M, Ely EW; MENDS investigators. Effect of dexmedetomidine versus lorazepam on outcome in patients with sepsis: an a priori-designed analysis of the MENDS randomized controlled trial. Crit Care. 2010;14(2):R38. doi: 10.1186/cc8916. Epub 2010 Mar 16. PMID 20233428
- [Background] Inouye SK. Delirium in older persons. N Engl J Med. 2006 Mar 16;354(11):1157-65. doi: 10.1056/NEJMra052321. No abstract available. PMID 16540616
- [Background] Pandharipande PP, Pun BT, Herr DL, Maze M, Girard TD, Miller RR, Shintani AK, Thompson JL, Jackson JC, Deppen SA, Stiles RA, Dittus RS, Bernard GR, Ely EW. Effect of sedation with dexmedetomidine vs lorazepam on acute brain dysfunction in mechanically ventilated patients: the MENDS randomized controlled trial. JAMA. 2007 Dec 12;298(22):2644-53. doi: 10.1001/jama.298.22.2644. PMID 18073360
- [Background] Schoenfeld DA, Bernard GR; ARDS Network. Statistical evaluation of ventilator-free days as an efficacy measure in clinical trials of treatments for acute respiratory distress syndrome. Crit Care Med. 2002 Aug;30(8):1772-7. doi: 10.1097/00003246-200208000-00016. PMID 12163791
- [Background] Riker RR, Shehabi Y, Bokesch PM, Ceraso D, Wisemandle W, Koura F, Whitten P, Margolis BD, Byrne DW, Ely EW, Rocha MG; SEDCOM (Safety and Efficacy of Dexmedetomidine Compared With Midazolam) Study Group. Dexmedetomidine vs midazolam for sedation of critically ill patients: a randomized trial. JAMA. 2009 Feb 4;301(5):489-99. doi: 10.1001/jama.2009.56. Epub 2009 Feb 2. PMID 19188334
- [Derived] Mistraletti G, Umbrello M, Salini S, Cadringher P, Formenti P, Chiumello D, Villa C, Russo R, Francesconi S, Valdambrini F, Bellani G, Palo A, Riccardi F, Ferretti E, Festa M, Gado AM, Taverna M, Pinna C, Barbiero A, Ferrari PA, Iapichino G; SedaEN investigators. Enteral versus intravenous approach for the sedation of critically ill patients: a randomized and controlled trial. Crit Care. 2019 Jan 7;23(1):3. doi: 10.1186/s13054-018-2280-x. PMID 30616675
- [Derived] Mistraletti G, Mantovani ES, Cadringher P, Cerri B, Corbella D, Umbrello M, Anania S, Andrighi E, Barello S, Di Carlo A, Martinetti F, Formenti P, Spanu P, Iapichino G; SedaEN investigators. Enteral vs. intravenous ICU sedation management: study protocol for a randomized controlled trial. Trials. 2013 Apr 3;14:92. doi: 10.1186/1745-6215-14-92. PMID 23551983